CLINICAL TRIAL: NCT05033093
Title: Effect of Resin, Calcium Silicate and Silicone Based Root Canal Sealers on Postoperative Pain: A Randomized Controlled Clinical Study
Brief Title: Effect of Resin, Calcium Silicate and Silicone Based Root Canal Sealers on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Esin Özlek, Asist. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/29.04.2021
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain
Keywords: root canal; root canal sealer; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Root Canal Filling Materials

STUDY DESIGN:
Intervention Model Description: After the final irrigation process root canals will be dried with sterile paper points and then randomly divided into three main groups according to the root canal sealer ; G1: AH Plus G2: iRoot SP G3: GuttaFlow Bioseal to be used in the obturation process (n: 28).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ah Plus (Active Comparator): All samples will be filled with Ah Plus root canal sealer and gutta percha
  Interventions: Drug: Root Canal Sealants
- I Root SP (Active Comparator): All samples will be filled with I Root SP root canal sealer and gutta percha
  Interventions: Drug: Root Canal Sealants
- GuttaFlow Bioseal (Active Comparator): All samples will be filled with GuttaFlow Bioseal canal sealer and gutta percha
  Interventions: Drug: Root Canal Sealants

INTERVENTIONS:
Drug: Root Canal Sealants — it is planned to conduct the research described below, on the effect of calcium silicate-based (iRoot SP), silicone-based (GuttaFlow Bioseal) and rezin-based (AH Plus) sealer on postoperative pain

SUMMARY:
After endodontic procedures, depending on the individual and many variables, postoperative pain can be occur within hours and continue for days following the treatment. It is thought that acute inflammation that develops due to chemical, mechanical or microbial injuries in the periapical tissue after endodontic treatment causes postoperative pain. Materials used for root canal obturation can reach periodontal tissues through the apical foramen, lateral canals or leakage and may affect the healing process in the periodontium. For this reason, knowing the properties of root canal obturation materials is important in terms of preventing postoperative pain.

Calcium silicate-based root canal sealer are recommended to be used as they enhance healing after endodontic treatment by promoting differentiation of odontoblasts and the release of bioactive compounds. At the same time, it has been reported that it has less cytotoxic effect compared to the resin-based AH Plus, which is widely used for root canal). Silicone-based root canal sealers have good biological properties on human ligament periodontal fibroblasts. It has been reported that GuttaFlow Bioseal root canal sealer, which has been used in recent years, has less cytotoxic effect than GuttaFlow2, MTA Fillapex and AH Plus sealers. Ateş et al.(2019) evaluated that the effects of different root canal sealers on postoperative pain and reported that the use of iRoot SP or AH Plus did not significantly affect pain levels, but iRoot SP sealer required less analgesic intake than AH Plus sealer. Aslan et al. (2020) concluded in their study that calcium silicate and resin-based root canal sealers are similar in terms of postoperative pain and need for analgesic intake. Ferreira et al.(2020) compared the effects of AH Plus, Endofill and MTA Fillapex root canal sealers on postoperative pain and stated that all three root canal sealers cause similar pain levels.

When reviewing the studies on postoperative pain, it is seen that mostly resin and calcium silicate based root canal sealers are evaluated. Studies on calcium silicate and silicone-based root canal sealers seem to focus more on cytotoxicity. However, no study has been found in the literature on the effect of GuttaFlow Bioseal sealer on postoperative pain, which has been popularity in recent years and has low cytotoxicity. Acoording to this information, it is planned to conduct the research described below, on the effect of calcium silicate-based (iRoot SP), silicone-based (GuttaFlow Bioseal) and rezin-based (AH Plus) sealer on postoperative pain.

DETAILED DESCRIPTION:
The study is planned to be carried out on 84 patients who were diagnosed and followed up in Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Endodontics, aged between 18-50 years, without any systemic disease. Patients diagnosed with irreversible pulpitis will be included in the study group. Patients with periapical lesions and open apex teeth will not be included in the study group. Before the treatment, pain levels of patients will be record according to the VAS scale.

Dental anesthesia will be achieved using local anesthetic solution (Maxicaine DS fort, Vem, Istanbul, Turkey) for inferior alveolar nerve blockade. After rubber dam isolation, endodontic access cavity will be prepared using high-speed burs. The working length will be determined with using apex locator (Propex Pixi, Dentsply Maillefer) and periapical radiographs with placing a #15 K-file (VDW GmbH, Munich, Germany) into the root canals at the end of the apical narrowing. The root canals will be mechanically prepared using ProTaperNext (DentsplyMaillefer,Baillagues,Switzerland) up to the X3 numbered instrument as standard in each patient. During instrumentation, irrigation will be performed with 2 mL 5.25% NaOCl (Microvem AF, İstanbul, Türkey) at each file change. A dental injector and a 27 gauge dental needle tip will be used for irrigation. The tip of the cannulas will be adjusted to reach two-thirds of the working size. According to the final irrigation procedure, all canals will be irrigated with 5 mL of 17% EDTA solution (Imicryl, Konya, Turkey), 5 mL of 5.25% NaOCI solution and 5 mL of saline, respectively.

After the final irrigation process root canals will be dried with sterile paper points and then randomly divided into three main groups according to the root canal sealer (G1: AH Plus; G2: iRoot SP; G3: GuttaFlow Bioseal) to be used in the obturation process (n: 28). All groups will be filled with sterile gutta-percha and root canal sealers in the same session using the single-cone technique. Teeth with completed root canal treatment will be restored with coronal sealing. After the treatment, patients in all three groups will be asked to report their pain levels according to the VAS scale at certain intervals (6th hour - 24th hour - 48. hour - 72. hour - 1st week) and their need of analgesic use. According to the questionnaires collected with patient feedback, pain levels will be evaluated after root canal treatment completed in a single session.

Descriptive statistics in terms of the features emphasized; It will be expressed as Average, Standard Deviation, Minimum and Maximum value. In order to compare the groups and Times (6, 24, 48, 72nd Hour and 1st Week) in terms of these characteristics, directional analysis of variance with two factors and one factor repeated, will be used. Duncan test will be used to identify different groups following analysis of variance. In determining the relationship between these variables, Pearson correlation coefficients will be calculated separately for the groups. Statistical significance level will be taken as 5% in calculations and SPSS statistical package program will be used for calculations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 45 years
* Mandibular molar teeth that were diagnosed with symptomatic irreversible pulpitis

Exclusion Criteria:

* Patients who are taken analgesic inflammatory drugs with in the last 12 hours
* Pregnancy or lactation
* Teeth with calcified canals
* Teeth with periodontal diseases
* Teeth with sensitive to percussion and palpation
* Teeth with root resorption
* Teeth with immature/open apex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
VAS Scala | up to 7 days
  PP will be assessed with a VAS after endodontic treatment. The VAS consisted of a 100-mm hor- izontal ruler with marks every 10 mm and no numbers except a 0 at the first part of the scale and a 10 in the last part of the scale.

IPD SHARING:
Plan to Share IPD: No
After the final irrigation process root canals will be dried with sterile paper points and then randomly divided into three main groups according to the root canal sealer (G1: AH Plus; G2: iRoot SP; G3: GuttaFlow Bioseal) to be used in the obturation process (n: 28). All groups will be filled with sterile gutta-percha and root canal sealers in the same session using the single-cone technique. Teeth with completed root canal treatment will be restored with coronal sealing. After the treatment, patients in all three groups will be asked to report their pain levels according to the VAS scale at certain intervals (6th hour - 24th hour - 48. hour - 72. hour - 1st week) and their need of analgesic use. According to the questionnaires collected with patient feedback, pain levels will be evaluated after root canal treatment completed in a single session.

REFERENCES:
- [Background] Graunaite I, Skucaite N, Lodiene G, Agentiene I, Machiulskiene V. Effect of Resin-based and Bioceramic Root Canal Sealers on Postoperative Pain: A Split-mouth Randomized Controlled Trial. J Endod. 2018 May;44(5):689-693. doi: 10.1016/j.joen.2018.02.010. Epub 2018 Mar 20. PMID 29571915